CLINICAL TRIAL: NCT00340340
Title: Genetic Epidemiology of Lung Cancer and Smoking; Current Title: Environmental And Genetic Lung Cancer Etiology (EAGLE)
Brief Title: Genetic Epidemiology of Lung Cancer and Smoking
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901211; 01-C-N211
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
Keywords: Population-Based Case Control Study; Lung Cancer; Epidemiology; Smoking; Smokers; Genetics
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Newly diagnosed lung cancer cases
- Controls: Population-based controls

SUMMARY:
We will conduct an interdisciplinary case-control/sib-pair study of lung cancer designed to explore the genetic determinants both of lung cancer and of smoking. The study includes biospecimen collection as well as exposure information with power to address main genetic effects and gene-environment interactions.

This is an integrated proposal designed to address two major issues: the genetic determinants of lung cancer in smokers and the genetic determinants of smoking. Other important issues will be addressed in the study with a marginal additional cost to the main design. The study achieves excellent power for studying the main effects of genetic factors that are relatively common and good power for formal tests of interactive effects.

Using a case-control design, with questionnaire, medical record abstraction, and blood collection, we will investigate: main effects of genes on lung cancer risk; gene-environment and gene-gene effects in lung cancer etiology; gene effects on smoking persistence; gene effects on ever-never smoking; gene-psychological interactions in smoking behaviors.

In addition, we will collect viable lymphocytes from all study subjects and tumor, metaplastic and normal tissue samples from 100 surgical cases. With these data and tissues, we will be able to study: genetic instabilities in lung cancer tissue in relation to specific exposures, genotype, persistence of smoking, and clinical presentation of lung cancer; histologic characteristics of lung cancer in relation to genotype, gene expression, somatic mutations, and smoking; functional assays in viable lmphocytes in relation to genotype, gene expression.

Finally, we will identify lung cancer-affected siblings of cases, and the unaffected siblings in the same sibships. This sample will permit us to: replicate associations found in the case-control sample with an alternative analytical method based on transmission statistics; address some population stratification issues.

DETAILED DESCRIPTION:
This is an interdisciplinary multicenter case-control study of lung cancer situated in Milan Italy, designed to explore the genetic determinants both of lung cancer and of smoking. We enrolled newly diagnosed lung cancer cases within a defined area around Milan Italy, and population-based controls from the same area. The study includes biospecimen collection as well as epidemiological and clinical data.

This is an integrated proposal designed to address two major issues: the genetic determinants of lung cancer and the genetic determinants of smoking. Other important issues arc addressed in the study with a marginal additional cost to the main design. The study achieves excellent power for studying the main effects of genetic factors that are relatively common and good power for formal tests of interactive eftects.

Using a case-control design, with questionnaire, medical record abstraction, and blood collection. we can investigate:

* main effects of genes on lung cancer risk
* gene-environment and gene-gene effects in lung cancer etiology
* gene effects on smoking persistence
* genes effects on ever-never smoking

In addition, we have collected viable lymphocytes from all study subjects and tumor, metaplastic and normal tissue samples from at least 400 surgical cases. With these data and tissues, we can study:

* genetic instabilities in lung cancer tissue in relation to specific exposures, genotype, persistence of smoking, and clinical presentation of lung cancer;
* histologic characteristics of lung cancer in relation to genotype, gene expression, methylation. somatic mutations, and smoking;
* functional assays in viable lymphocytes in relation to genotype, gene expression

Moreover. we are collecting clinical reports of treatments, quality of life, recurrence, toxicities, and survival from all cases that consented. With this material we will be able to link the genetic profiles of the cases with data on therapy efficacy, toxicity and survival, to contribute to the improvement of treatment for lung cancer.

ELIGIBILITY:
* INCLUSION CRITERIA - CASE GROUP:

The case group will consist of 2,000 newly incident lung cancer cases, male and female, 35 to 79 years old, with verified lung cancer, collected before or after surgery and prior to chemotherapy or radiation therapy.

All histologic types and all stages of lung cancer will be eligible.

Cases will be consecutively collected in the departments of thoracic surgery, general surgery, general medicine, and oncology.

The pool of cases will be residents of Lombardy derived from 5 cities (Milan, Brescia, Varese, Monza, and Pavia) and the surrounding residential villages served by 14 hospitals, that encompass all five medical schools in the region.

Enrolled cases will have no history of other cancers, except for basal cell carcinoma of the skin or in situ cervical carcinoma.

Subjects in intensive care units, or with cardiac, hepatic, renal, or CNS failure, or with uncompensated schizophrenia, psychosis, or inability to speak, will not be enrolled.

All subjects will sign an informed consent.

INCLUSION CRITERIA - CONTROL GROUP:

The control group will consist of 2,000 gender-, age-, and county-matched controls with no history of cancer.

We will choose a population-based or hospital-based control group depending on the result of a pilot study.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer cases consecutively enrolled from 13 hospitals and population-based controls with no cancer.
Sampling Method: Probability Sample
Enrollment: 4429 (Actual)
Dates: Start 2001-06-28 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Tobacco smoking and other exposures and genetic susceptibility measures | Ongoing
  Risk of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Landi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (18):
- Italy (18):
  - Ospedale Fatebenefratelli Sant'Orsola, Brescia
  - Spedali Civili, Brescia
  - Azienda Ospedaliera San Paolo, Milan
  - Euromedia Marketing Service, Milan
  - Fondazione Centro San Raffaele - HSR, Milan
  - Hosp Niguarda Ca Granda, Milan
  - Istituti Clinici de Perfezionamento ICP, Milan
  - L'Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Ospedale Maggiore di Milano, Milan
  - Ospedale San Carlo Borromeo, Milan
  - Ospedale San Giuseppe, Milan
  - Universita Degli Studi di Milano, Milan
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Interfield, Milan
  - Azienda Ospedaliera San Gerardo, Monza-Milano
  - Policlinico San Matteo, Pavia
  - Instituto Clinica Humanitas - ICH, Rozzano-Milan
  - Azienda Ospedale di Circolo di Varese, Varese

REFERENCES:
- [Background] Zuber V, Marconett CN, Shi J, Hua X, Wheeler W, Yang C, Song L, Dale AM, Laplana M, Risch A, Witoelar A, Thompson WK, Schork AJ, Bettella F, Wang Y, Djurovic S, Zhou B, Borok Z, van der Heijden HF, de Graaf J, Swinkels D, Aben KK, McKay J, Hung RJ, Bikeboller H, Stevens VL, Albanes D, Caporaso NE, Han Y, Wei Y, Panadero MA, Mayordomo JI, Christiani DC, Kiemeney L, Andreassen OA, Houlston R, Amos CI, Chatterjee N, Laird-Offringa IA, Mills IG, Landi MT. Pleiotropic Analysis of Lung Cancer and Blood Triglycerides. J Natl Cancer Inst. 2016 Aug 26;108(12):djw167. doi: 10.1093/jnci/djw167. Print 2016 Dec. PMID 27565901
- [Background] Yu G, Gail MH, Consonni D, Carugno M, Humphrys M, Pesatori AC, Caporaso NE, Goedert JJ, Ravel J, Landi MT. Characterizing human lung tissue microbiota and its relationship to epidemiological and clinical features. Genome Biol. 2016 Jul 28;17(1):163. doi: 10.1186/s13059-016-1021-1. PMID 27468850
- [Background] Shi J, Hua X, Zhu B, Ravichandran S, Wang M, Nguyen C, Brodie SA, Palleschi A, Alloisio M, Pariscenti G, Jones K, Zhou W, Bouk AJ, Boland J, Hicks B, Risch A, Bennett H, Luke BT, Song L, Duan J, Liu P, Kohno T, Chen Q, Meerzaman D, Marconett C, Laird-Offringa I, Mills I, Caporaso NE, Gail MH, Pesatori AC, Consonni D, Bertazzi PA, Chanock SJ, Landi MT. Somatic Genomics and Clinical Features of Lung Adenocarcinoma: A Retrospective Study. PLoS Med. 2016 Dec 6;13(12):e1002162. doi: 10.1371/journal.pmed.1002162. eCollection 2016 Dec. PMID 27923066